CLINICAL TRIAL: NCT04370327
Title: The Effects of Claudication Severity on Functional Outcomes in Patients With Intermittent Claudication
Brief Title: The Effects of Claudication Severity on Functional Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Stefan Birkett, Lecturer In Exercise Science, University of Central Lancashire
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UCentalLancashirePAD
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Free Exercise (PF) (Active Comparator): Patients will be randomised to twice weekly for 24 weeks of pain free exercise in a supervised exercise programme
  Interventions: Other: Pain Free Exercise (PF)
- Moderate Claudication Pain Exercise (MOD-P) (Active Comparator): Patients will be randomised to twice weekly for 24 weeks of moderate claudication pain exercise in a supervised exercise programme
  Interventions: Other: Moderate Claudication Pain Exercise (MOD-P)
- Maximal Claudication Pain Exercise (MAX-P) (Active Comparator): Patients will be randomised to twice weekly for 24 weeks of maximal claudication pain exercise in a supervised exercise programme
  Interventions: Other: Maximal Claudication Pain Exercise (MAX-P)

INTERVENTIONS:
Other: Pain Free Exercise (PF) — Patients will exercise until the onset on claudication (1 on the rating scale)
  Arms: Pain Free Exercise (PF)
Other: Moderate Claudication Pain Exercise (MOD-P) — Patients will exercise until they experience moderate claudication pain (2 on the rating scale)
  Arms: Moderate Claudication Pain Exercise (MOD-P)
Other: Maximal Claudication Pain Exercise (MAX-P) — Patients will exercise until they experience maximal claudication pain (4 on the rating scale)
  Arms: Maximal Claudication Pain Exercise (MAX-P)

SUMMARY:
Peripheral artery disease (PAD) affects over 236 million people globally. A classic symptom of PAD is intermittent claudication (IC) which is associated with reductions in physical function. The evidence is irrefutable that supervised exercise programmes (SEP) improve pain free and maximal waking distance. However, adherence rates are poor with exercise-related pain cited as contributable factor. Exercise at mild claudication or pain- free exercise improves walking ability, however current guidelines recommend exercise should be performed to near maximal claudication to improve walking ability. Conflicting evidence exists and there is a lack of evidence that has directly compared the relative effects of exercise prescribed at different levels of claudication. Therefore, the primary objective is to directly compare the effects of exercise prescribed at different levels of claudication pain on functional outcomes

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a progressive disease and is characterised by atherosclerotic occlusion of the arteries in the lower limbs, resulting in a reduction of blow flow. Globally, it is estimated that 236 million people are living with PAD, with the number of cases increasing by 24% from 2000 to 2010 (Song et al., 2019). A classic symptom of PAD is intermittent claudication (IC), which is characterised by ischemic muscle pain precipitated by exertion and relieved by rest. IC is associated with various comorbidities such as diabetes mellitus, hypertension and dyslipidaemia as well as reductions in physical function, quality of life, and balance. National and international guidelines recommend exercise therapy as first line treatment for patients with IC, advocating two hours per week of a supervised exercise over a three-month period, with patients being encouraged to exercise to the point of maximal pain. Exercise therapy is also a cost-effective option, as a three month programme costs less than a tenth of the cost of angioplasty.

However, despite the plethora of evidence demonstrating the benefits of SEP, less than half of vascular units in the United Kingdom (UK) have access one and patient uptake rates low. A lack of motivation has been shown as one of the primary reasons for poor adherence with claudication pain being suggested as a contributable factor. Indeed, exercise-induced pain has been shown as a major barrier to physical activity in this population and the level of pain prescribed during SEP influences completion rates. When exercise is prescribed at higher levels of pain, completion rates are lower. However, current evidence and guidelines advocate exercising to the point of near maximal pain, despite evidence to the contrary, suggesting that mild- or pain-free exercise improves walking ability. As such, it remains unclear which level of claudication is optimal for improving functional outcomes in patients with IC which can affect patient adherence, clinical practice and exercise prescription. The lack of adequately powered, randomised clinical trials investigating the effects of exercise prescribed at differing levels of claudication pain has also been highlighted in a recent scientific statement from the American Heart Association

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Resting ankle brachial pressure index (ABPI) <90 mmHg
3. Able to walk unaided
4. English speaking and able to follow exercise instructions
5. Able to provide informed consent

Exclusion Criteria:

1. Those who have critical limb threatening ischaemia (rest pain and/or tissue loss)
2. Unable to provide consent
3. Those undergoing active cancer treatment
4. Those presenting with any significant comorbidities or contraindications to exercise testing or training in accordance to the American College of Sports Medicine
5. Unstable/uncontrolled coronary heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Walking Distance (MWD) | 12 and 24 weeks
  Metres walked until maximal claudication pain

SECONDARY OUTCOMES:
Change in Pain Free Walking Distance (PFWD) | 12 and 24 weeks
  Metres walked pain free
Adherence | 24 weeks
  Recording the number of training sessions attended and successfully completed
Change in Quality of Life | 12 and 24 weeks
  King College 24-item Vascular Quality of life and walking impairment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Birkett, PHD, Principal Investigator — University of Central Lancashire
Locations (1):
- School of Sport and and Health Sciences, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birkett ST, Sinclair J, Seed SA, Pymer S, Caldow E, Ingle L, Harwood AE, Egun A. Effects of exercise prescribed at different levels of claudication pain on walking performance in patients with intermittent claudication: a protocol for a randomised controlled trial. Ther Adv Cardiovasc Dis. 2022 Jan-Dec;16:17539447221108817. doi: 10.1177/17539447221108817. PMID 35762773